CLINICAL TRIAL: NCT06373302
Title: Peripheral Arterial Disease Biomarkers: The Effect of Intervention on Biomarker Levels and Predictors of Restenosis or Deterioration
Brief Title: Peripheral Arterial Disease Biomarkers
Acronym: PADBIRD
Status: Not yet recruiting | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 323948
Record Dates: First submitted 2023-12-11; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral; Arterial; Disease; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercise Therapy: Patients who are advised by their clinician to undertake exercise therapy as their treatment for peripheral arterial disease
- Angioplasty: Patients undergoing angioplasty for treatment of peripheral arterial disease, as advised by their clinician.

SUMMARY:
The study aims to determine how expression levels of biomarkers for peripheral arterial disease change over time in response to exercise therapy, surgical or endovascular intervention, and whether they can be used to predict disease progression.

DETAILED DESCRIPTION:
Several studies have identified markers in the blood (called biomarkers) that are associated with peripheral arterial disease, or clogging up of the blood supply to the leg. There is little understanding however regarding how these respond to intervention, and how they are related to walking distance.

This study will increase the understanding of the relationship between peripheral arterial disease state and biomarker expression and enable us to work towards the development of new targets for treatment.

Participants will be invited to undertake questionnaires and dedicated walking tests alongside regular blood tests to check their biomarker levels. These will be undertaken on a regular basis so the investigators can see what happens over time, such as after a surgical procedure, and see if these markers go back towards normal following intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 50 years
* Symptomatic PAD
* ABPI <0.8 or TBPI <0.7

Exclusion Criteria:

* Aged <50 years
* Current Malignancy
* Rheumatological Condition
* Previous surgical or endovascular intervention for PAD
* ABPI >0.8 or TBPI >0.7

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between PAD biomarker levels and walking distance. | Baseline
  The correlation between PAD biomarker levels and walking distance.
Change in PAD biomarker levels following exercise therapy. | 6 months up to 2 years
  To investigate the change in PAD biomarker levels following exercise therapy.
Change in PAD biomarker levels following endovascular intervention | 48 hours
  To investigate the change in PAD biomarker levels following endovascular intervention

SECONDARY OUTCOMES:
To determine whether biomarker levels normalise with improved walking distance. | 2 years
  Change in biomarker levels in participants with improved walking distance compared to particicpants with static or deteriorating walking distance at 6 months.
To determine whether biomarker levels can be used as a predictor of restenosis, occlusion or reintervention following endovascular intervention. | 2 years
  Compare the change in biomarkers levels pre and post angioplasty between participants requiring reintervention or occlusion, and those not requiring re-intervention or occlusion.
Levels of biomarkers and (Major Adverse Cardiovascular Events). | 2 years
  The association between levels of biomarkers and (Major Adverse Cardiovascular Events).

IPD SHARING:
Plan to Share IPD: No